CLINICAL TRIAL: NCT04328038
Title: Personalized Exercise Oncology (PEXO) - Study
Brief Title: Personalized Exercise Oncology
Acronym: PEXO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Joachim Wiskemann, Head of Exercise Onoclogy, Principal Investigator, Associated Professor, University Hospital Heidelberg
Other Study IDs: HRP-591-PEXO
Record Dates: First submitted 2020-03-24; First posted 2020-03-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Health Behavior
Keywords: Physical Activity; Exercise; Health literacy; cancer-related symptoms; treatment-related symptoms; personalized Medicine
MeSH Terms: conditions — Neoplasms; Health Behavior; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- USA: Cohort from the USA
  Interventions: Other: Survey
- Germany: Cohort from Germany
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patient fill out a survey containing: Demographic Information, medical history, several Questionnaires about Health Literacy, Well Being/HRQoL and Fatigue

SUMMARY:
The Goal of the study is to identify trait-homogenous groups of cancer patients in regards to their physical activity associated health literacy. Based on these Groups, individualized exercise protocols and educative strategies can be developed which may increase the efficacy of the exercise therapy and increases the likelihood that patient get involved in physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer diagnosis
* Females and males ≥18 years of age
* Undergoing either chemo-, immune-, radio- or anti-hormonal treatment
* Last surgery more than 6 weeks in the past
* Ability to understand English or German
* Be able to provide and understand informed consent
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Score of ≤ 2

Exclusion Criteria:

* Heart insufficiency > NYHA III (New York Heart Association) or uncertain arrhythmia
* Uncontrolled hypertension
* Severe renal dysfunction (GFR < 30%, Creatinine> 3mg/dl)
* Reduced standing or walking
* Current pregnancy
* Any other evidence in the medical record of an absolute contraindication for exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mixed Cohort of adult cancer patients undergoing treatment Special Subgroup: Multiple Myeloma Patients
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Patient Clusters | through study completion, an average of 1 year
  Identification of different, trait-homogenous patient clusters

SECONDARY OUTCOMES:
Questionnaire: Physical Activity Associated Health Literacy | through study completion, an average of 1 year
  To assess physical activity-associated health competence the recently developed and validated questionnaire from Sudeck and Pfeifer (2016) will be used
Questionnaire: Health Literacy | through study completion, an average of 1 year
  To assess health-literacy the recently developed and validated questionnaire from Sudeck and Pfeifer (2016) will be used
Questionnaire: Health Related Quality of Life | through study completion, an average of 1 year
  Quality of Life will be assessed with the validated 30-item self-assessment questionnaire of the European Organization for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0).
Questionnaire: Fatigue | through study completion, an average of 1 year
  To asses fatigue patients will be asked to complete the 12-item EORTC QLQ-FA12 (FA = fatigue), which is a newly developed questionnaire which has been intensively validated
Questionnaire: Physical Activity | through study completion, an average of 1 year
  Patient's level of physical activity will be assessed with the SQUASH Physical Activity Questionnaire. It includes multiple activities referring to a 'normal' week. Activity dimensions asked include actively commuting physical activity (walking, cycling), physical activity at work or school, household activities, leisure time activities (sports, walking, gardening, cycling).
Questionnaire: Emotion Thermometers | through study completion, an average of 1 year
  Emotion thermometers are four-domain visual-analogue scale including distress, anxiety, depression, and anger. Each domain is rated on an 11-point (0 to 10) Likert scale
Questionnaire: Brief Pain Inventory (BPI) | through study completion, an average of 1 year
  Bone pain will be assessed with the Brief Pain Inventory (BPI). This is a valid and reliable tool for pain measurement in cancer patients with bone metastases. It measures both pain severity and pain interference on function

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg University Hospital, Heidelberg, Germany

REFERENCES:
- [Derived] Greinacher A, Kuehl R, Mai EK, Goldschmidt H, Wiskemann J, Fleischer A, Rasche L, Dapunt U, Maatouk I. The impact of divergent forms of social support on health-related quality of life in patients with multiple myeloma and its precursor states. J Cancer Res Clin Oncol. 2024 Jan 31;150(2):55. doi: 10.1007/s00432-023-05570-9. PMID 38291214
- [Derived] Kuehl R, Koeppel M, Goldschmidt H, Maatouk I, Rosenberger F, Wiskemann J. Physical activity-related health competence and symptom burden for exercise prescription in patients with multiple myeloma: a latent profile analysis. Ann Hematol. 2023 Nov;102(11):3091-3102. doi: 10.1007/s00277-023-05326-y. Epub 2023 Jun 24. PMID 37355476